CLINICAL TRIAL: NCT01775163
Title: E-MECHANIC Ancillary Study: Effect of Exercise-Induced Weight Loss on Energy Metabolism
Brief Title: Effect of Exercise-Induced Weight Loss on Energy Metabolism
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Leanne Redman, Principal Investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 10008-A
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Metabolism; Weight Loss
Keywords: Energy; Metabolism; Weight Loss; Exercise
MeSH Terms: conditions — Weight Loss; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Self Directed Exercise: Participants randomized to the self-directed group will receive information on physical activity recommendations and guidelines on nutrition aimed at promoting weight loss. Participants will not be given a specific exercise recommendation in terms of weekly energy expenditure.
- Low Intensity Exercise: Individuals assigned to the low dose exercise group will be required to expend 8 calories per kg of body weight per week in structured aerobic exercise on a treadmill or stationary bicycle. The exercise intensity will be maintained at 65% of VO2peak. The caloric goal of each session will be calculated by dividing the weekly caloric expenditure goal by participant selected exercise frequency (i.e., 3, 4 or 5 times per week). The training program consists of a 3-min warm-up at a progressively increasing intensity until the prescribed training intensity is reached. All exercise sessions are conducted at the PBRC Fitness Center and will be supervised by staff trained on the aspects of the study protocol.
- High Intensity Exercise: Individuals assigned to the low dose exercise group will be required to expend 20 calories per kg of body weight per week in structured aerobic exercise on a treadmill or stationary bicycle. The exercise intensity will be maintained at 65% of VO2peak. The caloric goal of each session will be calculated by dividing the weekly caloric expenditure goal by participant selected exercise frequency (i.e., 3, 4 or 5 times per week). The training program consists of a 3-min warm-up at a progressively increasing intensity until the prescribed training intensity is reached. All exercise sessions are conducted at the PBRC Fitness Center and will be supervised by staff trained on the aspects of the study protocol.

SUMMARY:
The E-MECHANIC Ancillary Study will measure changes in 24-hour energy expenditure and spontaneous physical activity in a subset of 60 obese individuals enrolled in the main study. We aim to determine if changes in energy metabolism might explain why people don't lose the expected amount of weight in an exercise program.

DETAILED DESCRIPTION:
This is an ancillary study to E-Mechanic, which is an National Institutes of Health study in 198 individuals with the objective to understand why certain people fail to lose weight in exercise programs. In E-Mechanic changes in body weight, body composition, energy intake and energy expenditure are measured before and after 3 different exercise programs of 24 weeks in duration. The 3 exercise programs being compared are self-directed exercise, low dose exercise and high dose exercise. The goal of this ancillary study is to undertake comprehensive assessments of energy metabolism in a metabolic chamber in a group of 60 obese individuals enrolled in the main study. We will compare differences in the changes in 24h energy expenditure and spontaneous physical activity between the 3 exercise programs. We will also test if changes in energy metabolism might explain why people don't lose the expected amount of weight after 24 weeks of exercise.

ELIGIBILITY:
Inclusion Criteria:

* Individuals enrolled in the E-MECHANIC main study (NCT#01264406) with a body mass index (BMI) greater than or equal to 30 kg/m2.

Exclusion Criteria:

* Not enrolled in the E-MECHANIC main study (NCT#01264406).
* Have a body mass index (BMI) less than 30 kg/m2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and Women enrolled in E-MECHANIC
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2010-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in 24h energy expenditure | 24 weeks
  24h energy expenditure will be measured in a room calorimeter before and after a 24 week exercise program

SECONDARY OUTCOMES:
Metabolic adaptation in 24h energy expenditure | 24 weeks
  The difference between the actual change in 24 energy expenditure and the energy expenditure estimated on the basis of body size will be compared between: 1) exercise groups and 2) between individuals who lost the expected amount of weight and individuals who did not lose the expected amount of weight during the exercise program

OTHER OUTCOMES:
Sleeping energy expenditure | 24 weeks
  Sleeping energy expenditure will be measured in a room calorimeter before and after a 24 week exercise program
Spontaneous physical activity | 24 weeks
  Spontaneous physical activity will be measured in a room calorimeter before and after a 24 week exercise program

CONTACTS AND LOCATIONS:
Overall Officials: Leanne M Redman, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Lam YY, Redman LM, Smith SR, Bray GA, Greenway FL, Johannsen D, Ravussin E. Determinants of sedentary 24-h energy expenditure: equations for energy prescription and adjustment in a respiratory chamber. Am J Clin Nutr. 2014 Apr;99(4):834-42. doi: 10.3945/ajcn.113.079566. Epub 2014 Feb 5. PMID 24500151